CLINICAL TRIAL: NCT01657929
Title: A Phase 1, Randomized Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of the H5-VLP + GLA-AF Pandemic Influenza Vaccine in Healthy Adult Subjects
Brief Title: H5-VLP + GLA-AF Vaccine Trial in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Collaborators: Medicago (Industry); Defense Advanced Research Projects Agency (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: IDRI-FPVPX-112
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Influenza A Subtype H5N1 Infection
Keywords: Influenza; Avian; H5N1; H5-VLP; GLA; GLA-AF
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 20 µg H5-VLP + 2.5 µg GLA-AF given ID (Experimental)
  Interventions: Biological: H5-VLP + GLA-AF
- 20 µg H5-VLP + 2.5 µg GLA-AF given IM (Experimental)
  Interventions: Biological: H5-VLP + GLA-AF
- 20 µg H5-VLP alone given ID (Active Comparator)
  Interventions: Biological: H5-VLP alone
- 20 µg H5-VLP + 1 mg Alhydrogel(R) given IM (Active Comparator)
  Interventions: Biological: H5-VLP + Alhydrogel(R)
- 90 µg licensed H5N1 vaccine (Active Comparator)
  Interventions: Biological: Licensed H5N1 vaccine

INTERVENTIONS:
Biological: H5-VLP + GLA-AF — H5-VLP antigen and GLA-AF adjuvant. 2 injections at Days 0, and 21.
  Arms: 20 µg H5-VLP + 2.5 µg GLA-AF given ID; 20 µg H5-VLP + 2.5 µg GLA-AF given IM
Biological: H5-VLP alone — H5-VLP antigen alone. 2 injections at Days 0, and 21.
  Arms: 20 µg H5-VLP alone given ID
Biological: H5-VLP + Alhydrogel(R) — H5-VLP antigen and Alhydrogel(R) adjuvant. 2 injections at Days 0, and 21.
  Arms: 20 µg H5-VLP + 1 mg Alhydrogel(R) given IM
Biological: Licensed H5N1 vaccine — Licensed H5N1 vaccine. 2 injections given on Days 0 and 21.
  Arms: 90 µg licensed H5N1 vaccine

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and immunogenicity in healthy adult subjects of an investigational vaccine being developed for the prevention of pandemic influenza. The vaccine, identified as H5-VLP + GLA-AF, consists of a recombinant influenza virus H5 protein (hemagglutinin from A/Indonesia/5/2005) produced in a plant-based expression system assembling into virus-like particles together with the adjuvant GLA-AF.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 49 years of age.
* Must be in good general health as confirmed by a medical history and physical exam, vital signs, and screening laboratories conducted no more than 30 days prior to study injection administration.
* Female subjects of childbearing potential, regardless of birth control history, must have a negative serum pregnancy test at screening, a negative urine pregnancy test on the day of each study injection, must not be breast-feeding or lactating, and are required to consistently use one of the following methods of contraception through the first three months of the study: hormonal (e.g. oral, transdermal, intravaginal, implant, or injection); double barrier (i.e., condom, diaphragm with spermicide); intrauterine device (IUD) or system (IUS); vasectomized partner (6 months minimum); abstinence (as confirmed by the investigator); or bilateral tubal ligation (if no conception post-procedure). These precautions are necessary due to unknown effects that H5-VLP + GLA AF or H5-VLP alone might have in a fetus or newborn infant. The subject must have no plan to become pregnant during the first three months of the study period. Females who are post-menopausal (no spotting at all) for at least one (1) year will not require a pregnancy test.
* The following screening laboratory blood tests must have values within the normal ranges (as provided by each clinical site) or not clinically significant as determined by the Principal Investigator (or designated sub-investigator) and Medical Monitor (all test results must be within 30 days prior to first study injection): sodium, potassium, BUN, ALT, AST, total bilirubin, alkaline phosphatase, creatinine, fasting glucose, fasting lipid panel, total WBC count, hemoglobin, and platelet count.
* The following serology tests must be negative: HIV 1/2 antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody.
* Negative urine test for recreational drugs and alcohol per Clinical Research Unit standards.
* Urinalysis not clinically significant as determined by the study clinician.
* In the opinion of the Investigator, must show comprehension of the study requirements, competence and willingness to provide written, informed consent for participation after reading the informed consent form. The subject must have adequate opportunity to discuss the study with an Investigator or qualified designee.
* Must be capable of completing a study memory aid in English.
* Must be able and willing to attend all evaluation visits, be reachable by telephone on a consistent basis by the study site personnel, and have a permanent address.

Exclusion Criteria:

* Previous exposure to H5N1 vaccines or experimental products containing GLA-AF.
* History of allergy to any of the constituents of H5-VLP (H5N1) + Alhydrogel (aluminum hydroxide) vaccine.
* Participation in another experimental protocol or receipt of any investigational or non-registered products within the past 3 months or planned use during the study period. Subjects may not participate in any other drug study while participating in this study.
* Treatment with immunosuppressive drugs (e.g., oral or injected steroids, such as prednisone; high dose inhaled steroids) or cytotoxic therapies (e.g., chemotherapy drugs or radiation) within the past 6 months.
* Received a blood transfusion or immunoglobulin within the past 3 months.
* Donated blood products (platelets, whole blood, plasma, etc.) within past 1 month.
* Poor venous access.
* Administration of any vaccine (including any other influenza vaccine) within a 30 day period prior to study enrollment, or planned administration of any vaccines within the period from the first study injection up to blood sampling at Day 42 or within 30 days prior to blood sampling at Day 189. Immunization on an emergency basis of a tetanus and diphtheria toxoids adsorbed for adult use (Td) will be allowed provided the vaccine is not administered within two weeks prior to study injection administration. Receipt of any other emergency immunizations (e.g. rabies) will result in a case-by-case review of continued participation.
* History of autoimmune disease or other causes of immunosuppressive states.
* Any confirmed or suspected immunosuppressive condition or immunodeficiency including history of human immunodeficiency virus (HIV) infection or presence of lymphoproliferative disease.
* History or evidence of any acute or chronic illness (including cardiovascular, pulmonary, neurological, hepatic, rheumatic, hematological, metabolic, or renal disorders, controlled hypertension), or use of medication that, in the opinion of the Principal Investigator (or designated sub-investigator), may interfere with the evaluation of the safety or immunogenicity of the vaccine.
* Cancer or treatment for cancer within 3 years of study injection administration. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Persons with treated and uncomplicated basal cell carcinoma of the skin are eligible.
* Presence of significant acute or chronic, uncontrolled medical or neuropsychiatric illness. "Uncontrolled" is defined as:

  * Requiring a new medical or surgical treatment within one month prior to study vaccine administration
  * Requiring a change in medication dosage in one month prior to test article administration due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable subjects are acceptable), or
  * Hospitalization or an event fulfilling the definition of a serious adverse event within one month prior to test article administration
* Rash, tattoos or any other dermatological condition that could adversely affect the vaccine injection site or interfere with its evaluation.
* BMI <18 or >30 kg/m2.
* Hypertension (systolic ≥150 mmHg or diastolic ≥90 mmHg).
* Resting pulse rate <40 bpm or >100 bpm.
* Any medical or neuropsychiatric condition which, in the Investigator's opinion, would render the subject incompetent to provide informed consent or unable to provide valid safety observations and reporting.
* Known or suspected alcohol or drug abuse within the past 6 months.
* Chronic smoker (> 20 pack years).
* History of allergy to tobacco or eggs.
* Subjects with a history of previous anaphylaxis or severe allergic reaction to vaccines, or unknown allergens.
* Subjects who are unlikely to cooperate with the requirements of the study protocol.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing adverse events | 385 days
  To evaluate the safety and tolerability of 20 μg of H5-VLP together with 2.5 μg of GLA-AF compared to 20 µg of H5-VLP alone, 20 µg of H5-VLP with 1 mg Alhydrogel(R), or a licensed H5N1 vaccine following intramuscular or intradermal administration on Days 0 and 21. The safety assessments will be based on local and systemic reactions, including reported adverse events, changes in laboratory values, and changes in vital signs. The severity and relationship to treatment will be recorded for all adverse events.

SECONDARY OUTCOMES:
Immunogenicity | Days 0, 7, 10, 21, 28, 31, 42, and 189
  To assess the immunogenicity of H5-VLP + GLA-AF compared to H5-VLP alone, H5-VLP + Alhydrogel, or a licensed H5N1 vaccine following intramuscular or intradermal administration by evaluating humoral and cellular responses to H5-VLP at specified timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Piazza, MD, MPH, Study Director — Access to Advanced Health Institute (AAHI)
Locations (3):
- United States (3):
  - Covance, Inc., Daytona Beach, Florida
  - Covance, Inc., Dallas, Texas
  - Covance, Inc., Madison, Wisconsin